CLINICAL TRIAL: NCT02076503
Title: Pre-operative PET-MR of High Risk Prostate Cancer Patients for Assessment of Cancer Aggressiveness and Lymph Node Status
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other); Norwegian Cancer Society (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2013/1513
Record Dates: First submitted 2014-02-10; First posted 2014-03-03 (Estimated); Last update posted 2018-01-05 (Actual); Status verified 2018-01

CONDITIONS: Prostatic Neoplasms
Keywords: Neoplasm Staging; Positron-Emission Tomography; Magnetic Resonance Imaging; 1-amino-3-fluorocyclobutane-1-carboxylic acid
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PET-MR 18F-FACBC (Experimental)
  Interventions: Procedure: PET-MR 18f-FACBC; Procedure: histology (gold standard)

INTERVENTIONS:
Procedure: PET-MR 18f-FACBC
Procedure: histology (gold standard) — histopathological classification of co-located dissected lymph nodes

SUMMARY:
Prostate cancer is the most frequent cancer in Norwegian men. For optimal treatment, accurate staging of the disease at the time point of diagnosis is important. The objective of this study is to evaluate the diagnostic potential of a combined PET/MR examination for risk assessment and detection of lymph node metastases. The overall aim of the project is to improve the investigators ability to provide individually tailored treatment to prostate cancer patients.

The study will include 32 men with high-risk prostate cancer, who are eligible for radical prostatectomy. Informed consent is a requirement for inclusion in the study.

ELIGIBILITY:
Inclusion Criteria:

* High-risk prostate cancer according to EAU guidelines (Gleason score ≥8 and/or PSA ≥20 ng/ml and/or ≥ cT3a cancer)
* Eligibility for the surgical procedure (radical prostatectomy and bilateral pelvic lymph node resection)

Exclusion Criteria:

* Previous treatment (for example TURP or hormone therapy)
* Contraindication for the PET/MR examination (including, but not limited to: pacemaker, aneurysm clips, reduced renal function, metal implants, claustrophobia)

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Positive and negative predictive value of 18FACBC PET/MR for detection of lymph node metastases | 7 days
  Findings on 18FACBC PET/MR images will be compared to histopathology, which is considered the gold standard for evaluation of pelvic lymph node metastases

CONTACTS AND LOCATIONS:
Overall Officials: Anders Angelsen, prof, Study Director — St. Olavs Hospital
Locations (1):
- Dept Urologic Surgery, St Olavs Hospital, Trondheim, Norway

REFERENCES:
- [Result] Elschot M, Selnaes KM, Sandsmark E, Kruger-Stokke B, Storkersen O, Tessem MB, Moestue SA, Bertilsson H, Bathen TF. A PET/MRI study towards finding the optimal [18F]Fluciclovine PET protocol for detection and characterisation of primary prostate cancer. Eur J Nucl Med Mol Imaging. 2017 Apr;44(4):695-703. doi: 10.1007/s00259-016-3562-7. Epub 2016 Nov 5. PMID 27817158
- [Result] Selnaes KM, Kruger-Stokke B, Elschot M, Willoch F, Storkersen O, Sandsmark E, Moestue SA, Tessem MB, Halvorsen D, Kjobli E, Angelsen A, Langorgen S, Bertilsson H, Bathen TF. 18F-Fluciclovine PET/MRI for preoperative lymph node staging in high-risk prostate cancer patients. Eur Radiol. 2018 Aug;28(8):3151-3159. doi: 10.1007/s00330-017-5213-1. Epub 2018 Jan 2. PMID 29294158